CLINICAL TRIAL: NCT02791295
Title: Diet and Physical Activity Lifestyle Intervention to Prevent Body Weight Gain in Patients With Type 2 Diabetes Starting Insulin Pump Treatment: a Randomized Controlled Trial
Brief Title: Lifestyle Intervention in Type 2 Diabetes
Acronym: WeightPump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icadom (Industry)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A00481-50
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes; lifestyle intervention; insulin pump treatment; body weight; body composition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body Weight | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet and physical activity program (Experimental): Diet and physical activity program with individual coaching
  Interventions: Other: Diet and physical activity program
- control (No Intervention): standard care

INTERVENTIONS:
Other: Diet and physical activity program — A personalized intervention focused on improving diet and increasing physical activity will be implemented at-home with a monthly support by a registered dietician and physical activity educator during 6 months
  Arms: Diet and physical activity program

SUMMARY:
The purpose of the study is to determine whether a personalized lifestyle intervention focused on diet and physical activity reinforcement is effective in avoiding weight gain in the first months following initiation of subcutaneous insulin pump therapy in type-2 diabetic patients.

DETAILED DESCRIPTION:
Patients with type 2 diabetes using insulin pump therapy are gaining weight within the first months of treatment. This weight gain could counterbalance the metabolic benefice of insulin pump treatment in improving glycemic control and could lead to treatment dropout. Lifestyle intervention aiming at improving physical activity and diet in type 2 diabetes is known to brought body weight reduction and cardiometabolic improvement.

The investigator hypothesized that an intensive, home-based, 6-months diet and physical activity program could prevent the body weight gain associated with insulin pump treatment initiation. The investigator will randomize patients with type 2 diabetes into a "lifestyle intervention" arm or a "usual care" control arm at the time of insulin pump treatment initiation. The primary objective will evaluate body weight change at 6 months after insulin pump treatment initiation. The secondary objectives will evaluate change in glycemic control (HbA1c) and body composition at 6 months. In addition, the retention effect will be assessed on body weight change one year after insulin pump treatment initiation, 6 months after the end of the lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult Type 2 diabetic patients with indication of initiation of insulin pump therapy.
* Patients addressed for the insulin pump follow-up to the home care provider supporting the study.
* Public health care security affiliation.

Exclusion Criteria:

* Breastfeeding or pregnant woman.
* Not willing to participate as assessed by the investigator.
* Patient engaged in another clinical trial with exclusion criteria for other protocol.
* Patients unable to ride a training bike.
* Unavailable in the next 6 months.
* Patient without a medical certificate done in the last 12 months by a cardiologist attesting the ability to participate in a physical activity reinforcement program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Weight change | 6 months
  The difference in body weight changes between the two groups over a six-month period following initiation of insulin pump treatment.

SECONDARY OUTCOMES:
Glycemic control | 6 months
  The difference in HbA1c changes between the two groups after 6-months of insulin pump treatment initiation.
Body composition | 6 months
  The difference between the two groups in distribution of fat mass and lean mass between the first visit and 6 months after initiation of insulin pump treatment.
Diabetes Treatment Satisfaction | 6 months
  The difference between the two groups of scores of the Diabetes Treatment Satisfaction Questionnaire between the first visit and 6 months after initiation of insulin pump treatment.
Intermediate weight change | 3 months
  The difference in weight changes between the two groups after 3-months of insulin pump treatment initiation.
Retention of weight change | 1 year
  The difference in weight changes between the two groups at 12-months of insulin pump treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Borel, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (6):
- France (6):
  - Annecy-Genevois Hospital, Annecy
  - Pierre Oudot Hospital, Bourgoin
  - Métropole Savoie Hospital, Chambéry
  - Alpes Léman Hospital, Contamine-sur-Arve
  - Grenoble University Hospital, Grenoble
  - Marseille European Hospital, Marseille

IPD SHARING:
Plan to Share IPD: No